CLINICAL TRIAL: NCT04707820
Title: Antiviral T Lymphocyte Immunity During Acute COVID-19 Infection
Acronym: ImmuCoV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/0100/HP
Record Dates: First submitted 2020-12-29; First posted 2021-01-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Enzyme-Linked Immunospot Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): - Patient with an acute SARS-CoV-2 infection, confirmed by PCR or typical CT images, requiring hospitalization in a COVID unit at Rouen University Hospital.
  Interventions: Diagnostic Test: ELISPOT
- control group (No Intervention): - Rouen University Hospital staff free of any symptomatology compatible with an SARS-CoV-2 infection (fever, cough, fatigue, loss of taste, loss of smell) since February 1, 2020

INTERVENTIONS:
Diagnostic Test: ELISPOT — The evolution of the number of gamma interferon (IFN) producing T lymphocytes in response to Spike glycoprotein (Spike glycoprotein) will be assessed by enumeration in ELISPOT method at 4 measurement times: D0 (confirmation of infection by PCR), D+7, D+14 or at hospital departure (D+Departure) and D+56±14 days.
  The ELISPOT method consists in stimulating peripheral blood mononuclear cells (isolated by density gradient and containing a known CD3+ T lymphocyte count) over a short period of time (16 to 20 hours) with a pool of 15 amino acid peptides (overlapping on 11 amino acids) representative of the S protein.
  Arms: Patient group

SUMMARY:
The SARS-CoV-2 (COVID-19) infection is causing a global pandemic and a major health crisis in France.

Immunity is the body's ability to defend itself against infectious agents such as viruses. The progressive acquisition by a large part of the population of immunity to defend itself against the COVID-19 virus is one of the main mechanisms by which a resolution of this pandemic is hoped for. Recovery from infection and protection from the virus is likely to depend on the development of antibodies (proteins produced by the body to neutralize infectious agents) and T-cells (a type of white blood cell in the immune system) that can stop the virus from multiplying and killing it.

To date, the way and speed at which the T-lymphocytes active against the virus appear are not known. The development of biological tests to detect T-cells active against the virus in the blood of infected patients is therefore necessary.

In this context, we propose you to participate in a study that will study the immune system's response against the sars-CoV-2 virus during and after COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an acute SARS-CoV-2 infection, confirmed by PCR or typical CT images, requiring hospitalization in a COVID unit at the Rouen University Hospital (pneumonic form requiring oxygen therapy < 4 L/min.)
* Rouen University Hospital staff free of any symptomatology compatible with an SARS-CoV-2 infection (fever, cough, fatigue, loss of taste, loss of smell) since February 1, 2020
* Age ≥ 18 years old
* Adult patient who has read and understood the information letter and signed the consent form
* Affiliation to a social security scheme

Exclusion Criteria:

* Patient with PCR-confirmed SARS-CoV-2 infection and hospitalized in intensive care units (acute respiratory distress and/or organ failure, whose pathogenesis may differ from the more frequently described forms with secondary aggravation (5)).
* Patient with PCR-confirmed but non-hospitalized SARS-CoV-2 infection (non-acute form, managed by confinement)
* A person participating in a therapeutic trial that may interfere with the procedures being investigated, including lymphocyte response prior to D+56±14 days.
* Known Pregnancy
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection / subtutorship or guardianship
* Staff at the Rouen University Hospital with SARS-CoV-2 infection confirmed by PCR and/or typical scan images during the epidemic period.
* Hospital staff who were exposed to the virus (working in a Covid unit)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Evolution of the number of gamma interferon (IFN) producing T lymphocytes in response to the S protein | for 56 days
  The evolution of the number of interferon-gamma producing T lymphocytes (IFN) in response to protein S (Spike glycoprotein) will be assessed by enumeration in ELISPOT method

SECONDARY OUTCOMES:
Numbers of T lymphocytes producing IFN in response to other CoV-2-SARS viral | for 56 days
  Numbers of T lymphocytes producing IFN in response to other CoV-2-SARS viral proteins (nucleoprotein, membrane proteins E (FEV1) and M (FEV1), proteins 3a, 9b, ORF10, non-structural proteins 6, 7a, 7b, 8, protein14) measured by ELISPOT
Anti-SARS-CoV-2 IgG and IgM levels | for 56 days
  Anti-SARS-CoV-2 IgG and IgM levels
SARS-CoV-2 viral load in nasopharyngeal swab | for 56 days
  SARS-CoV-2 viral load in nasopharyngeal swab

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France